CLINICAL TRIAL: NCT05363969
Title: Treatment of Self Harm Scars With Fraxel Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Darius Mehregan (Other)
Responsible Party: Sponsor-Investigator, Darius Mehregan, Chairman Dept of Dermatology, Wayne State University
Organization: Wayne State University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21-06-3672
Record Dates: First submitted 2022-04-21; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Self Harm
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fractionated laser resurfacing — Patients will receive 3-4 treatments with fractionated laser resurfacing
  Other Names: Fraxel

SUMMARY:
Treatment of self harm scars with fractionated laser.

DETAILED DESCRIPTION:
Fractionated resurfacing lasers have been shown to be useful for scars including acne scars, burns scars and striae. We will treat self harm scars with 3 to 4 treatments using a "Fraxel" fractionated laser. Patients will be screened to ensure they are not actively engaged in self harm behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Self harm scars

Exclusion Criteria:

* Active self harm behaviors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement of scars | 6 months
  Patients will be assessed with pre and post treatment photography. Photographs will be taken at baseline and 1 month after the final treatment. After the final treatment both the investigator and patients will rate appearance of scarring as "worsened", "unchanged" or "improved" as compared to baseline.

IPD SHARING:
Plan to Share IPD: No